CLINICAL TRIAL: NCT04316689
Title: Open-label, Phase 1 Study of S-488210/S-488211 to Evaluate the Safety and Tolerability in Patients With Unresectable Recurrent and/or Metastatic Solid Tumor
Brief Title: First-in-human Study of S-588210 (S-488210+S-488211)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1801P2011
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer; Head and Neck Cancer; Bladder Cancer; Esophageal Cancer; Mesothelioma
Keywords: Metastatic solid tumor; Unresectable recurrent solid tumor; S-588210; Peptide vaccine
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Mesothelioma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- S-588210 (S-488210 + S-488211) (Experimental): Participants will receive subcutaneous injections once a week for 4 weeks and then a biweekly extension treatment for 8 weeks. Each treatment will consist of 1 subcutaneous injection of 1 mL of S- 488210 and 1 subcutaneous injection of 1 mL of S-488211 containing 1 mg each of the 5 peptides.
  Interventions: Biological: S-488210; Biological: S-488211

INTERVENTIONS:
Biological: S-488210 — S-488210 is a freeze-dried injectable formulation containing the following three peptides, S-488201 (a URLC10-derived peptide), S-488202 (a CDCA1-derived peptide) and S-488203 (a KOC1-derived peptide).
  Other Names: S-588210
Biological: S-488211 — S-488211 is a freeze-dried injectable formulation containing the following two peptides, S-488204 (a DEPDC1-derived peptide) and S-488205 (an MPHOSPH1-derived peptide).
  Other Names: S-588210

SUMMARY:
The primary objective is to evaluate the safety and tolerability of S-588210 (S-488210+S-488211) in patients with unresectable recurrent and/or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable recurrent and/or metastatic solid tumor of lung, esophageal, head and neck, mesothelioma, or bladder cancer (including urothelial cancer of renal pelvis, ureters, and urethra), who have progressed after conventional systemic therapies or have exhausted or are intolerant to existing treatment options.
2. Human leukocyte antigen (HLA)-A*02:01-positive patients.
3. Patients who are male or female aged ≥18 years at the time of informed consent.
4. Patients with the Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1 at enrollment.
5. Patients who have a lymphocyte count accounting for 15% or higher of the total white blood cell count within 28 days before enrollment.
6. Patients who provide a personally signed and dated informed consent document for participation in the study.
7. Patients with expected life-span of at least 3 months from the time of enrollment.

Exclusion Criteria:

1. Patients who are expected to require any of the following therapies between enrollment and completion of the Observation Period.

   * Anti-malignant tumor drug
   * Systemic corticosteroid (except for corticosteroid defined as the equivalent of prednisone ≤ 10 mg/day orally)
   * Systemic immunosuppressant drug
   * Radiotherapy (except for restricted radiotherapy for pain relief of bone metastasis) for the cancer(s)
   * Surgical therapy for the cancer(s)
   * Hyperthermia for the cancer(s)
   * Traditional Chinese herbal medicine with anti-tumor or immunosuppressant effect
   * Other investigational products
2. Patients who have severe concurrent hepatic impairment, renal impairment, heart disease, hematological disease, respiratory disease, or metabolic disease, with the exception of any symptoms and/or signs associated with cancer(s).
3. Patients who have known human immunodeficiency virus infection.
4. Patients with uncontrolled systemic or active infection.
5. Patients who had any diseases with the risk of sudden death within 12 months before enrollment.
6. Patients with a history or evidence of autoimmune diseases and/or immunodeficiencies.
7. Female patients who are pregnant, breastfeeding, or have a positive pregnancy test at the predose examinations.
8. Patients who are considered ineligible for this study by the investigator or subinvestigator due to any reasons, including inability to understand and follow the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 16 weeks
  Adverse events will be classified by system organ class and preferred term using Medical Dictionary for Regulatory Activities (MedDRA).

SECONDARY OUTCOMES:
Cytotoxic T Lymphocyte (CTL) Induction Rate | Baseline and Weeks 8 and 12
  CTL induction is defined as the increase in CTL activity at any point after baseline. Accordingly, the CTL induction rate is calculated as the percentage of participants who show CTL induction to at least any of the 5 antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- University College London Clinical Research Facility, London, United Kingdom